CLINICAL TRIAL: NCT01305421
Title: The Role of the Grip Test in the Evaluation of Extubation Success in ICU Patients.
Brief Title: Grip Test in Ventilated ICU Patients
Acronym: griptest92
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Brugmann (Other)
Responsible Party: De Bels, David, MD, CHU Brugmann
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: griptest92
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Mechanically Ventilated ICU Patients
Keywords: ICU; muscle strength; mechanical ventilation; weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: grip test — Muscle strength measurement by hand-held dynamometer

SUMMARY:
ICU patients do experience extubation failure. Guidelines rarely include muscle strength criteria. Prior work indicates that grip strength is a reliable surrogate for muscle strength. The purpose of the study is to assess the success rate of mechanical ventilation weaning based on the grip test.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated ICU patients

Exclusion Criteria:

* tracheotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Extubation success | 48 hours without reintubation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium